CLINICAL TRIAL: NCT05757544
Title: A Study to Optimize the Dosing Regimen and Assess Safety and Efficacy of IV Ganaxolone as Adjuvant Therapy for Established Status Epilepticus
Brief Title: Safety and Efficacy Study of IV Ganaxolone as Adjuvant Therapy for Established Status Epilepticus (ESE)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: for business reasons
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1042-SE-2002
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Status Epilepticus
Keywords: Established status epilepticus; Ganaxolone; Antiepileptic drug; Adjuvant therapy
MeSH Terms: conditions — Status Epilepticus | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participating staff involved in the evaluation and execution of the study will remain blinded to the participant's treatment assignment during the double-blind phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose optimization phase (open label): IV Ganaxolone bolus (variable) followed by infusion (variable) (Experimental)
  Interventions: Drug: IV Ganaxolone
- Double-blind phase: IV Ganaxolone + SOC (Experimental)
  Interventions: Drug: IV Ganaxolone
- Double-blind phase: IV Placebo + SOC (Placebo Comparator)
  Interventions: Drug: IV Placebo

INTERVENTIONS:
Drug: IV Ganaxolone — IV Ganaxolone will be administered.
  Arms: Dose optimization phase (open label): IV Ganaxolone bolus (variable) followed by infusion (variable); Double-blind phase: IV Ganaxolone + SOC
Drug: IV Placebo — IV Placebo will be administered
  Arms: Double-blind phase: IV Placebo + SOC

SUMMARY:
This study is designed to optimize the dosing regimen and evaluate the preliminary safety and efficacy of Intravenous (IV) ganaxolone as adjuvant therapy for participants with ESE receiving initial IV antiepileptic drug (AED) according to currently practiced standard of care (SOC). The study will be composed of 2 phases: an initial, open-label, dose optimization phase followed by IV ganaxolone versus placebo double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age at the time of the first IP bolus dose.
2. Has received benzodiazepines before or after arrival to the ED for generalized convulsive seizures lasting more than 5 minutes.
3. Has received the last dose of benzodiazepine more than 5 minutes prior to the first IP bolus initiation.
4. Ongoing or recurrent convulsions, or evidence of electrographic SE on rapid EEG immediately prior to the first IP bolus initiation.
5. The participant has not yet received a second-line IV AED for the treatment of the current episode of SE or the first IP bolus can be initiated within 15 minutes before or 10 minutes after the administration of such IV AED(s).

Exclusion Criteria:

1. The participant is intubated or the decision to proceed with intubation has been made.
2. The cause of SE is acute anoxic brain injury, cardiac arrest, acute trauma, hyper- or hypo-glycemia, or eclampsia.
3. The participant is known or suspected to be pregnant.
4. The participant is incarcerated at the time of SE occurrence.
5. Participants who pre-emptively opted out of the study.
6. A known allergy or sensitivity to progesterone or allopregnanolone medications/ supplements.
7. Receiving a concomitant IV product containing Captisol®.
8. Known estimated glomerular filtration rate (eGFR) <30 milliliters per minute (mL/min) and not receiving dialysis (may initiate first IP bolus prior to acute labs).
9. Individual weighing or suspected to weigh <40 kilograms (kg).
10. Hypotension requiring 2 or more vasopressors.
11. An individual who, in the opinion of the investigator has a life expectancy of less than 24 hours.
12. Use of an investigational product for which less than 30 days or 5 half-lives have elapsed from the final product administration. Participation in a non-interventional clinical study does not exclude eligibility.
13. Known or suspected history or evidence of a medical condition that, in the investigator's judgment, would expose participant to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Absence of electrographic (rapid electroencephalography [EEG]) evidence of status epilepticus or recurrence of convulsions at 1 hour after the first IP bolus administration without the use of any additional medications with anti-seizure properties | At 1 hour

SECONDARY OUTCOMES:
Percentage of participants with no escalation of care for Status epilepticus (SE) during investigational product (IP) infusion | Up to Day 7
Time to clinical seizure and electrographic SE cessation | Up to Day 7
Percentage of participants with no escalation of care (including re-administration of IP) at any point within 24 hours from the initial IP bolus administration | Up to 24 hours
Percentage of participants with no escalation to IV anesthesia for treatment of seizures during IP infusion | Up to Day 7
Percentage of participants with no escalation to IV anesthesia for treatment of seizures within 24 hours of the initial IP bolus | Up to 24 hours
Time to clinical or electrographic seizure recurrence within 24 hours from the initiation of the first IP bolus | Up to 24 hours

IPD SHARING:
Plan to Share IPD: No